CLINICAL TRIAL: NCT01816074
Title: Sequencing Treatments for Mothers With ADHD and Their At - Risk Children
Acronym: TMF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Mark Stein, Professor/Director, Seattle Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-0189
Record Dates: First submitted 2013-03-05; First posted 2013-03-21 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Mothers; ADHD; Treatment; Child
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Maternal Medication then meds (Experimental): The mothers in this treatment arm are given an active medication to treat ADHD (Vyvanse) in the first phase of the study, and in the second phase are randomized to enhanced medication
  Interventions: Drug: Vyvanse (lisdexamphetamine)
- BPT then continued beh tx (Experimental): The mothers in this treatment arm are given Behavior Parent Training in the first phase of the study, and in the second phase are randomized to enhanced behavioral treatment.
  Interventions: Behavioral: Behavior Parent Training
- Maternal Medication then BPT (Experimental): The mothers in this treatment arm are given an active medication to treat ADHD (Vyvanse) in the first phase of the study, and in the second phase are randomized to combined treatment (adding Behavior Parent Training).
  Interventions: Drug: Vyvanse (lisdexamphetamine); Behavioral: Behavior Parent Training
- BPT then maternal medication (Experimental): The mothers in this treatment arm are given Behavior Parent Training in the first phase of the study, and in the second phase are randomized to active ADHD medication, Vyvanse.
  Interventions: Drug: Vyvanse (lisdexamphetamine); Behavioral: Behavior Parent Training

INTERVENTIONS:
Drug: Vyvanse (lisdexamphetamine) — Active ADHD drug, Vyvanse, is administered to mother.
  Other Names: Lisdexamfetamine
  Arms: BPT then maternal medication; Maternal Medication then BPT; Maternal Medication then meds
Behavioral: Behavior Parent Training — Mother is given 8 weeks of individual sessions of behavioral parent training
  Other Names: BPT
  Arms: BPT then continued beh tx; BPT then maternal medication; Maternal Medication then BPT

SUMMARY:
We hypothesize that successfully treating maternal Attention Deficit Hyperactivity Disorder (ADHD) will have a beneficial effect that extends to the child. We believe that multi-component interventions combining maternal stimulant medication, Lisdexamfetamine (LDX), and Behavioral Parent Training (BPT) will improve parenting, maternal, and child outcomes. In terms of improved parenting, we hypothesize that some mothers may respond well to LDX or BPT alone and therefore may not require multi-modal treatment, whereas others may benefit most from multi-modal treatment

DETAILED DESCRIPTION:
The overarching goal of this study is to construct and evaluate an adaptive intervention (i.e., an individualized treatment protocol that is adjusted based on the child-mother dyad's initial response to treatment) to improve the trajectory of ADHD outcomes in at-risk children. Our primary outcome measure for the child will be whether child ADHD symptoms on the Conners Parent and Teacher Rating Scales decreased at the completion of the study. Our secondary outcome measure will be whether there was a need for medication for the child over the course of the study. The primary outcome for the mother will be the Conners Adult ADHD Rating Scale (CAARS) Attention Scale and the Clinical Global Impression-Severity scale (CGI-S).

ELIGIBILITY:
Mothers Inclusion Criteria:

* Sign informed consent
* Be between 21-50 years old (inclusive) at the screening visit and English-speaking
* At screening (after washout, if required) meet full Diagnostic and Statistical Manual (DSM-IV) criteria for ADHD, any subtype
* Have current CGI-S-ADHD rating > 4 and < 8
* Have findings on physical exam (PE), laboratory studies, vital signs, and electrocardiogram (ECG) judged to be normal for age with no contraindications for methylphenidate (MPH) treatment
* Have pulse and blood pressure (BP) within 95% of age and gender mean
* Commit to the entire visit schedule for the study
* Be able to complete all study assessments
* Women of childbearing potential (not surgically sterile or post-menopausal) must agree to use a medically-accepted contraception method consistently
* Mothers with comorbid mood/anxiety disorders which are effectively treated with Selective Serotonin Reuptake Inhibitors (SSRIs) will be eligible for participation, provided this medication has not changed within 30 days, is well tolerated, and that current mood symptoms are not severe or associated with active suicidal ideation. Also, the prescribing physician must approve of their participation in the study.

Mothers Exclusion Criteria:

* History of allergic reactions or severe negative response to study medications
* History of alcohol/substance abuse in the past 3 months or a positive urinary toxic screen on initial evaluation that is not explained by a time-limited medical circumstance
* History of or current bipolar illness, schizophrenia, psychoses, or significant suicidal risk
* History of chronic or acute medical disorder for which stimulant therapy would be contraindicated (e.g., glaucoma, hypertension)

Child Inclusion Criteria:

* Sign assent if older than 6
* Be between the ages of 4-8
* symptoms of ADHD (Conners Hyperactivity Index > 60), no prior treatment with effective doses of stimulants, defined as one or more weeks of treatment with adequate doses.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Stein, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Derived] Lui JHL, Chronis-Tuscano A, Almirall D, Whitlock KB, French W, Stein MA. Sequencing Stimulant Medication and Behavioral Parent Training in Multiplex ADHD Families: A Pilot SMART. J Clin Psychiatry. 2025 Feb 19;86(1):24m15463. doi: 10.4088/JCP.24m15463. PMID 40009046
- [Derived] Chronis-Tuscano A, French W, Strickland J, Sasser T, Gonzalez ENS, Whitlock KB, Stein MA. Acute Effects of Parent Stimulant Medication Versus Behavioral Parent Training on Mothers' ADHD, Parenting Behavior, and At-Risk Children. J Clin Psychiatry. 2020 Sep 8;81(5):19m13173. doi: 10.4088/JCP.19m13173. PMID 32926603

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited from the investigators' practices, clinic referrals, online advertisements, and radio advertisements. Participants were enrolled between September 2012 and December 2016.
Pre-assignment Details: 7 participants didn't meet inclusion criteria, 1 decided not to participate after screening, 2 withdrew due to time commitment issues, 1 had a comorbid psychiatric disorder, 1 had a physical contraindication.
Groups:
- Maternal Medication Then Additional Maternal Medication: The mothers in this treatment arm are given an active medication to treat ADHD (Vyvanse) in the first phase of the study, and in the second phase are randomized to enhanced medication
  Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother.
- Maternal Behavioral Parent Training (BPT) Then Additional BPT: The mothers in this treatment arm are given Behavior Parent Training in the first phase of the study, and in the second phase are randomized to enhanced behavioral treatment.
  Behavior Parent Training: Mother is given 8 weeks of individual sessions of behavioral parent training
Period: Phase 1
Arm/Group | Maternal Medication Then Additional Maternal Medication | Maternal Behavioral Parent Training (BPT) Then Additional BPT | Maternal Medication Then BPT | BPT Then Maternal Medication
Started | 11 | 9 | 11 | 10
Completed | 11 | 9 | 10 | 10
Not Completed | 0 | 0 | 1 | 0
Not completed — Time commitment issues | 0 | 0 | 1 | 0
Period: Phase 2
Arm/Group | Maternal Medication Then Additional Maternal Medication | Maternal Behavioral Parent Training (BPT) Then Additional BPT | Maternal Medication Then BPT | BPT Then Maternal Medication
Started | 11 | 9 | 10 | 10
Completed | 9 | 7 | 10 | 9
Not Completed | 2 | 2 | 0 | 1
Not completed — Time commitment Issues | 0 | 2 | 0 | 0
Not completed — Unsatisfied with Randomization assignmen | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: We enrolled a total of 53 mother-child dyads (total of 106 participants), 41 dyads were randomized to a treatment arm and completed the baseline visit (total of 82 participants). The number of participants in this section is double that of the participant flow because the dyads are split to accurately analyze characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maternal Medication Then Meds | BPT Then Continued Beh tx | Maternal Medication Then BPT | BPT Then Maternal Medication | Total
Number analyzed (Participants) | 22 | 18 | 22 | 20 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 41 dyads were randomized to treatment and completed a baseline visit. The dyads are separated to analyze the baseline characteristics: moms and children. This means that there are a total of 41 moms and 41 children for a total of 82 participants.
  years
    Mom age: number analyzed (Participants) | 11 | 9 | 11 | 10 | 41
    Mom age | 40.55 (7.31) | 39.00 (5.94) | 37.82 (5.78) | 41.00 (6.73) | 39.59 (6.38)
    Child age: number analyzed (Participants) | 11 | 9 | 11 | 10 | 41
    Child age | 6.00 (1.73) | 5.89 (1.05) | 6.18 (1.47) | 6.60 (1.35) | 6.17 (1.41)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: 41 dyads were randomized to treatment and completed a baseline visit. The dyads are separated to analyze the baseline characteristics: moms and children. This means that there are a total of 41 moms and 41 children for a total of 82 participants.
  Participants
    Child gender: number analyzed (Participants) | 11 | 9 | 11 | 10 | 41
    Child gender: Male | 6 | 6 | 6 | 5 | 23
    Child gender: Female | 5 | 3 | 5 | 5 | 18
    Parent gender: number analyzed (Participants) | 11 | 9 | 11 | 10 | 41
    Parent gender: Male | 0 | 0 | 0 | 0 | 0
    Parent gender: Female | 11 | 9 | 11 | 10 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 41 dyads were randomized to treatment and completed a baseline visit. The dyads are separated to analyze the baseline characteristics: moms and children. This means that there are a total of 41 moms and 41 children for a total of 82 participants.
  Participants
    Mom: number analyzed (Participants) | 11 | 9 | 11 | 10 | 41
    Mom: Hispanic or Latino | 2 | 0 | 1 | 1 | 4
    Mom: Not Hispanic or Latino | 9 | 9 | 10 | 9 | 37
    Mom: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
    Child: number analyzed (Participants) | 11 | 9 | 11 | 10 | 41
    Child: Hispanic or Latino | 0 | 0 | 2 | 1 | 3
    Child: Not Hispanic or Latino | 9 | 8 | 7 | 8 | 32
    Child: Unknown or Not Reported | 2 | 1 | 2 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 41 dyads were randomized to treatment and completed a baseline visit. The dyads are separated to analyze the baseline characteristics: moms and children. This means that there are a total of 41 moms and 41 children for a total of 82 participants.
  Participants
    Mother Race: number analyzed (Participants) | 11 | 9 | 11 | 10 | 41
    Mother Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Mother Race: Asian | 0 | 0 | 0 | 0 | 0
    Mother Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Mother Race: Black or African American | 1 | 0 | 0 | 1 | 2
    Mother Race: White | 9 | 9 | 9 | 7 | 34
    Mother Race: More than one race | 1 | 0 | 2 | 1 | 4
    Mother Race: Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
    Child Race: number analyzed (Participants) | 11 | 9 | 11 | 10 | 41
    Child Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Child Race: Asian | 0 | 0 | 0 | 0 | 0
    Child Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Child Race: Black or African American | 1 | 0 | 0 | 1 | 2
    Child Race: White | 9 | 9 | 9 | 8 | 35
    Child Race: More than one race | 0 | 0 | 2 | 1 | 3
    Child Race: Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Child Behavioral Functioning
Description: Child symptom severity will be assessed using the Clinical Global Impression - Severity (CGI-s) scale. This was collected at Baseline, Week 8 (end of Phase 1) and Week 16 (end of Phase 2). The CGI-S scale summarizes the clinician's impression of the participant's symptom improvement and ranges from 1-7 with 1 representing very much improved and 7 representing very much worse.
Time Frame: Baseline, Weeks 8 and 16
Population: 7 participants had missing data, the Child CGI-S was not collected at any of the study visits for these participants because they completed the study before this measure was added to the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Medication Then Additional Maternal Medication | Maternal Behavioral Parent Training (BPT) Then Additional BPT | Maternal Medication Then BPT | BPT Then Maternal Medication
Number analyzed (Participants) | 9 | 9 | 9 | 9
units on a scale
  Baseline | 4.78 (0.92) | 4.56 (1.42) | 4.44 (0.96) | 4.67 (1.33)
  Week 8 | 4.33 (0.67) | 3.75 (1.09) | 3.63 (0.99) | 3.78 (0.63)
  Week 16 | 4.13 (0.93) | 3.67 (1.25) | 3.38 (1.22) | 3.22 (0.92)

2. Secondary Outcome: Maternal Behavioral Functioning
Description: The Clinical Global Impression - Severity (CGI-S) scale will be used. This was collected at Baseline, Week 8 (end of Phase 1) and Week 16 (end of Phase 2). The CGI-S scale summarizes the clinician's impression of the participant's symptom improvement and ranges from 1-7 with 1 representing very much improved and 7 representing very much worse.
Time Frame: Baseline, Weeks 8 and 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maternal Medication Then Additional Maternal Medication | Maternal Behavioral Parent Training (BPT) Then Additional BPT | Maternal Medication Then BPT | BPT Then Maternal Medication
Number analyzed (Participants) | 11 | 11 | 11 | 10
units on a scale
  Baseline | 4.64 (0.64) | 4.50 (0.50) | 4.82 (0.72) | 4.45 (0.50)
  Week 8 | 3.55 (0.50) | 3.67 (0.67) | 2.60 (0.66) | 3.80 (0.87)
  Week 16 | 3.20 (0.60) | 3.86 (0.35) | 2.60 (1.02) | 2.56 (0.96)

3. Other Pre Specified Outcome: Parental and Family Functioning
Description: The Dyadic Parent-Child Interaction Coding System (DPICS) will be used at baseline, week 8, and week 16 to provide an observational measure of positive and negative behaviors of the mother toward the child. Instances of positive (e.g. praise) and negative (e.g. criticism) behaviors are coded by study raters trained to reliability; scores range from 0 to no upper limit. Higher numbers indicate higher instances of the observed behaviors.
Time Frame: Baseline, Weeks 8 and 16
Population: 6 participants were in the study before this assessment was added. 2 participants did not complete this assessment before they withdrew from the study. 3 participants withdrew from the study after the baseline visit (1 in the medication then medication arm after week 8, 1 in the Medication then BPT arm and 1 in BPT then BPT arm).
Measure: Mean (Standard Deviation); unit: instances observed
Groups:
- Maternal Medication Then Additional Maternal Med - Baseline; Maternal Medication Then Additional Maternal Med - Week 8; Maternal Medication Then Additional Maternal Med - Week 16: The mothers in this treatment arm are given an active medication to treat ADHD (Vyvanse) in the first phase of the study, and in the second phase are randomized to enhanced medication
  Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother.
- Maternal Medication Then Behavior Parent Training - Baseline; Maternal Medication Then Behavior Parent Training - Week 8; Maternal Medication Then Behavior Parent Training - Week 16: The mothers in this treatment arm are given an active medication to treat ADHD (Vyvanse) in the first phase of the study, and in the second phase are randomized to combined treatment (adding Behavior Parent Training).
  Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother.
  Behavior Parent Training: Mother is given 8 weeks of individual sessions of behavioral parent training
- Behavior Parent Training Then Maternal Medication - Baseline; Behavior Parent Training Then Maternal Medication - Week 8; Behavior Parent Training Then Maternal Medication - Week 16: The mothers in this treatment arm are given Behavior Parent Training in the first phase of the study, and in the second phase are randomized to active ADHD medication, Vyvanse.
  Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother.
  Behavior Parent Training: Mother is given 8 weeks of individual sessions of behavioral parent training
- Behavior Parent Training Then Additional BPT - Baseline; Behavior Parent Training Then Additional BPT - Week 8; Behavior Parent Training Then Additional BPT - Week 16: The mothers in this treatment arm are given Behavior Parent Training in the first phase of the study, and in the second phase are randomized to enhanced behavioral treatment.
  Behavior Parent Training: Mother is given 8 weeks of individual sessions of behavioral parent training
Arm/Group | Maternal Medication Then Additional Maternal Med - Baseline | Maternal Medication Then Additional Maternal Med - Week 8 | Maternal Medication Then Additional Maternal Med - Week 16 | Maternal Medication Then Behavior Parent Training - Baseline | Maternal Medication Then Behavior Parent Training - Week 8 | Maternal Medication Then Behavior Parent Training - Week 16 | Behavior Parent Training Then Maternal Medication - Baseline | Behavior Parent Training Then Maternal Medication - Week 8 | Behavior Parent Training Then Maternal Medication - Week 16 | Behavior Parent Training Then Additional BPT - Baseline | Behavior Parent Training Then Additional BPT - Week 8 | Behavior Parent Training Then Additional BPT - Week 16
Number analyzed (Participants) | 9 | 9 | 8 | 9 | 8 | 8 | 9 | 9 | 9 | 8 | 7 | 7
instances observed
  Total Positive Parenting | 23.61 (13.70) | 27.17 (12.39) | 32.56 (16.75) | 41.67 (26.03) | 31.55 (19.73) | 51.70 (25.04) | 21.83 (13.93) | 46.33 (28.65) | 44.07 (46.78) | 17.49 (10.48) | 34.71 (14.65) | 39.52 (20.06)
  Total Negative Parenting | 11.33 (11.36) | 17.01 (12.79) | 10.51 (10.80) | 8.64 (5.19) | 13.47 (14.58) | 5.96 (5.32) | 8.04 (6.77) | 5.01 (4.74) | 7.66 (6.64) | 10.64 (6.28) | 9.44 (4.48) | 8.85 (4.34)

ADVERSE EVENTS:
Time Frame: 16 weeks. Adverse events were collected from participants while they were in the study. Adverse events were not collected from participants that were not currently on medication including the BPT then BPT arm and the BPT then Medication arm while in the BPT phase.
Description: At each weekly visit, the parent met with the investigators and research staff. Investigators inquired about any side effects the parent experienced and recorded responses.
Groups:
- Vyvanse 20 mg: Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother. For the mothers that were randomized to medication arm, 20mg was the first dose they received.
- Vyvanse 30 mg: Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother. For the mothers that were randomized to medication arm, 30mg was offered to the mother if 20mg was not a strong enough dose.
- Vyvanse 40mg: Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother. For the mothers that were randomized to medication arm, 40mg was offered to the mother if 30mg was not a strong enough dose.
- Vyvanse 50 mg: Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother. For the mothers that were randomized to medication arm, 50mg was offered to the mother if 40mg was not a strong enough dose.
- Vyvanse 60 mg: Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother. For the mothers that were randomized to medication arm, 60mg was offered to the mother if 50mg was not a strong enough dose.
- Vyvanse 70mg: Vyvanse (lisdexamphetamine): Active ADHD drug, Vyvanse, is administered to mother. For the mothers that were randomized to medication arm, 70mg was offered to the mother if 60mg was not a strong enough dose.
Arm/Group | Vyvanse 20 mg | Vyvanse 30 mg | Vyvanse 40mg | Vyvanse 50 mg | Vyvanse 60 mg | Vyvanse 70mg
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/22 | 0/19 | 0/12 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 11/27 | 12/22 | 12/19 | 5/12 | 4/6 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vyvanse 20 mg (N=27) | Vyvanse 30 mg (N=22) | Vyvanse 40mg (N=19) | Vyvanse 50 mg (N=12) | Vyvanse 60 mg (N=6) | Vyvanse 70mg (N=2)
Appetite Suppression (Gastrointestinal disorders) | 5 (6) | 5 (9) | 3 (3) | 1 (3) | 3 (4) | 1 (2)
Irritability (General disorders) | 4 (4) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Sleep Disturbance or Fatigue (General disorders) | 6 (8) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Jitteriness/Restlessness (General disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Cardiac Events (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Includes events such as elevated BP, racing heart, thumping heart, etc.
Illness/Infection (General disorders) | 1 (1) | 6 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Includes colds, influenza, upper respiratory infection, urinary tract infection, etc.
Gastrointestinal issues (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Includes GI slowing, constipation, GERD, stomachaches
Headache (General disorders) | 2 (4) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hives (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Increased Menstraul Cramps (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diaphoresis (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tense (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scotomata (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No